CLINICAL TRIAL: NCT00511706
Title: Safety and Efficacy of a New Treatment as Adjunctive Therapy to Anti-vascular Endothelial Growth Factor (Anti-VEGF) Treatment in Patients With Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 206207-016
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Choroidal Neovascularization; Age-Related Maculopathy
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Dexamethasone; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone and ranibizumab (Experimental): Intravitreal injection of dexamethasone 700 µg at Day 1; ranibizumab 500 µg at Day -30 and Day 7-14.
  Interventions: Drug: dexamethasone; Biological: ranibizumab
- sham and ranibizumab (Sham Comparator): Sham injection at Day 1; ranibizumab 500 µg at day -30 and Day 7-14.
  Interventions: Biological: ranibizumab; Other: sham

INTERVENTIONS:
Drug: dexamethasone — Intravitreal injection of dexamethasone 700 µg at Day 1.
  Other Names: Posurdex
  Arms: dexamethasone and ranibizumab
Biological: ranibizumab — Ranibizumab 500 µg at day -30 and Day 7-14.
  Other Names: Lucentis®
Other: sham — Sham needle-less injection administered in the study eye at Day 1.
  Arms: sham and ranibizumab

SUMMARY:
The study will evaluate the safety and efficacy of the intravitreal implant of dexamethasone with Anti-VEGF treatment vs. Anti-VEGF alone (with sham dexamethasone injection) in patients with subfoveal choroidal neovascularization secondary to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older with subfoveal choroidal neovascularization (CNV) (classic and/or occult) secondary to AMD
* Visual Acuity between 20/40 and 20/400 in the study eye

Exclusion Criteria:

* Any intraocular surgery within 3 months
* Glaucoma
* Cataract
* High eye pressure
* Uncontrolled systemic disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2007-11-01 (Actual); Primary Completion 2009-03-01 (Actual); Study Completion 2009-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (9):
- Boynton Beach, Florida, United States
- Parramatta, New South Wales, Australia
- Paris, France
- Tel Aviv, Israel
- Milan, Italy
- Auckland, New Zealand
- Coimbra, Portugal
- Seoul, South Korea
- Southampton, Hampshire, United Kingdom

REFERENCES:
- [Background] Kuppermann BD, Goldstein M, Maturi RK, Pollack A, Singer M, Tufail A, Weinberger D, Li XY, Liu CC, Lou J, Whitcup SM; Ozurdex(R) ERIE Study Group. Dexamethasone Intravitreal Implant as Adjunctive Therapy to Ranibizumab in Neovascular Age-Related Macular Degeneration: A Multicenter Randomized Controlled Trial. Ophthalmologica. 2015;234(1):40-54. doi: 10.1159/000381865. Epub 2015 Jun 18. PMID 26088793

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone and Ranibizumab | Sham and Ranibizumab
Started | 123 | 120
Completed | 115 | 115
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone and Ranibizumab | Sham and Ranibizumab | Total
Number analyzed (Participants) | 123 | 120 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.1 (8.83) | 76.2 (8.50) | 76.1 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 69 | 145
  Male | 47 | 51 | 98

OUTCOME MEASURES:

1. Primary Outcome: Injection Free Interval
Description: The injection free interval was defined as the number of days between receiving the second ranibizumab injection (day 7 to 14) to the investigator's determination of eligibility to receive a third ranibizumab injection in the study eye.
Time Frame: Week 1 to Week 25
Population: Intent-to-treat population consisted of all randomized patients.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Dexamethasone and Ranibizumab | Sham and Ranibizumab
Number analyzed (Participants) | 123 | 120
Days | 34 [28 to 85] | 29 [28 to 56]

2. Secondary Outcome: Change From Baseline in the Best Corrected Visual Acuity (BCVA) at Week 25
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Baseline, Week 25
Population: Participants from the Intent-to-treat population (all randomized patients) with data available at Baseline and Week 25 for analyses.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Dexamethasone and Ranibizumab | Sham and Ranibizumab
Number analyzed (Participants) | 122 | 120
Letters
  Baseline | 55.5 (15.27) | 58.1 (12.64)
  Change from baseline at week 25 | 2.0 (8.61) | 2.4 (9.14)

3. Secondary Outcome: Change From Baseline in the Mean Central Retinal Subfield Thickness at Week 25 as Assessed by Optical Coherence Tomography (OCT) in the Study Eye
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina, was performed in the study eye after pupil dilation at baseline and Month 25.
Time Frame: Baseline, Week 25
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Dexamethasone and Ranibizumab | Sham and Ranibizumab
Number analyzed (Participants) | 120 | 119
Microns
  Baseline | 260.28 (123.625) | 272.45 (130.829)
  Change from baseline at week 25 (n=105, 111) | -7.12 (77.898) | -13.00 (97.651)

4. Secondary Outcome: Change From Screening in the Area of Leakage From Choroidal Neovascularization (CNV) at Week 25 as Assessed by Fluorescein Angiography in the Study Eye
Description: Fluorescein angiography (FA) is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Photographs are taken with a specialized low-power microscope with an attached camera designed to photograph the interior of the eye, including the retina and optic disc. FA was performed on the study eye after dilation at Screening and Week 25.
Time Frame: Screening (-Week 28), Week 25
Population: Participants from the intent-to-treat population (all randomized participants) with data available at Screening and Week 25 for analyses.
Measure: Mean (Standard Deviation); unit: Millimeters square (MM^2)
Arm/Group | Dexamethasone and Ranibizumab | Sham and Ranibizumab
Number analyzed (Participants) | 118 | 116
Millimeters square (MM^2)
  Screening | 8.44 (6.863) | 8.12 (6.359)
  Change from Screening at Week 25 (n= 95,99) | -2.32 (4.927) | -1.73 (5.465)

ADVERSE EVENTS:
Description: Safety population was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events and was defined as all randomized participants who received study drug.
Arm/Group | Dexamethasone and Ranibizumab | Sham and Ranibizumab
Serious Adverse Events (participants affected / at risk) | 9/121 | 14/118
Other Adverse Events (participants affected / at risk) | 86/121 | 59/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone and Ranibizumab (N=121) | Sham and Ranibizumab (N=118)
Renal failure (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0 — verbatim term= digoxin toxicity
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3
Myocardial infarction (Cardiac disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Stupor (Nervous system disorders) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Hernia (General disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone and Ranibizumab (N=121) | Sham and Ranibizumab (N=118)
Conjunctival haemorrhage (Eye disorders) | 23 | 12
Intraocular pressure increased (Eye disorders) | 16 | 5
Retinal haemorrhage (Eye disorders) | 9 | 7
Visual acuity reduced (Eye disorders) | 9 | 5
Macular degeneration (Eye disorders) | 6 | 5
Vitreous floaters (Eye disorders) | 6 | 2
Cataract subcapsular (Eye disorders) | 6 | 1
Eye pain (Eye disorders) | 5 | 8
Cataract (Eye disorders) | 4 | 7
Vitreous detachment (Eye disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.